CLINICAL TRIAL: NCT04205864
Title: Application of Thrombin Gel Matrix for the Prevention of Lymphocele in Patients With Endometrial Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KIA 2019/93
Record Dates: First submitted 2019-12-13; First posted 2019-12-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Lymphocele; Lymphocele After Surgical Procedure; Endometrium Cancer
MeSH Terms: conditions — Lymphocele; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: Application of Thrombin gel matrix after Pelvic lymphadenectomy. And compare this application with Conventional Pelvic Lymphadenectomy.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional pelvic lymphadenectomy (Active Comparator): Conventional pelvic lymphadenectomy
  Interventions: Procedure: Conventional Pelvic lymphadenectomy
- Thrombin gel matrix pelvic lymphadenectomy (Experimental): Thrombin gel matrix applicated after conventional pelvic lymphadenectomy
  Interventions: Drug: Thrombi-Gel

INTERVENTIONS:
Drug: Thrombi-Gel — Thrombin gel Matrix applied on pelvic lymphadenectomy areas after lympadenectomy
  Arms: Thrombin gel matrix pelvic lymphadenectomy
Procedure: Conventional Pelvic lymphadenectomy — Conventional Pelvic lymphadenectomy
  Arms: Conventional pelvic lymphadenectomy

SUMMARY:
To compare the incidence of lymphocele in Endometrial cancer patients with thrombin gel matrix used and not used during pelvic lymph node dissection.

DETAILED DESCRIPTION:
Pelvic lymph node dissection is the most accurate staging tool to determine lymph node involvement in endometrial cancer. Lymphoceles developed after surgery can cause serious morbidity, additional costs and delays in chemotherapy or radiotherapy. In this study, conventional pelvic lymphadenectomy will be compared with thrombin gel matrix application after pelvic lymphadenectomy. Our goal is to prospectively assess the lymphostatic effect of thrombin gel matrix in endometrial cancer patients undergoing pelvic lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer patients who need laparotomic bilateral PLND
* Patients suitable for surgery

Exclusion Criteria:

* Previous pelvic surgery
* Previous Chemotherapy or Radiotherapy
* Patients who undergo only lymph node sampling
* Patients who have not signed Informed Consent

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 72 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Frequency of pelvic lymphocele | post-operative 2th month
  Frequency pelvic lymphocele at post-operative 2th month

SECONDARY OUTCOMES:
Volume of radiographic lymphoceles | post-operative 2th month
  Volume of lymphocele detected with radiographic imagining at post-operative 2th month (the two largest dimensions measured in centimetres)
duration of postoperative drainage catheter | up to post-operative 1 week
  duration of postoperative drainage catheter
Postoperative drain amount (ml: milliliters) | with 1 weeks after surgery
  Postoperative drain amount (ml: milliliters)

CONTACTS AND LOCATIONS:
Overall Officials: Şener Gezer, M.D, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YH, Shin HJ, Ju W, Kim SC. Prevention of lymphocele by using gelatin-thrombin matrix as a tissue sealant after pelvic lymphadenectomy in patients with gynecologic cancers: a prospective randomized controlled study. J Gynecol Oncol. 2017 May;28(3):e37. doi: 10.3802/jgo.2017.28.e37. Epub 2017 Feb 28. PMID 28382800